CLINICAL TRIAL: NCT05162157
Title: Home Spirometry for the Diagnosis and Monitoring of Asthma and COPD in Primary Care in The Netherlands and Sweden: an Implementation Study
Brief Title: Home Spirometry in Primary Care: an Implementation Study
Acronym: Spiro@Home
Status: Completed | Type: Observational
Sponsor: General Practitioners Research Institute (Network)
Responsible Party: Sponsor
Other Study IDs: GPRI-21003-SPI
Record Dates: First submitted 2021-09-27; First posted 2021-12-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: COPD Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- at-home spirometry: This group performs spirometry at home with the Nuvoair spirometer
  Interventions: Device: NuvoAir platform

INTERVENTIONS:
Device: NuvoAir platform — Nuvoair platform, consisting of a bluetooth spirometer, smartphone application and clinical portal

SUMMARY:
Rationale: Spirometry is essential in the diagnosis of airway disease and can be useful in monitoring patients. Despite the essential role, spirometry remains largely underused in primary care. Due to Coronavirus disease (COVID-19), the use of office spirometry is contraindicated in many countries. Furthermore, spirometric devices are costly and personnel requires special training. Referral for spirometry increases the cost for patients and lowers the feasibility. Part of the reason for underdiagnosis of airway disease are the specific situations (such as exercise-induced asthma) in which spirometry in office setting might not reveal abnormalities. In recent years, handheld spirometry linked to phones/apps has been developed for study purposes and remote monitoring.

Objective: To study the feasibility, quality and added value of at-home spirometry for the diagnosis and monitoring of asthma and Chronic Obstructive Pulmonary Disease (COPD) in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Spirometry indication
* Able and willing to use at-home spirometry

Exclusion Criteria:

* On the discretion of the recruiting clinician if he or she deems a patient not eligible.
* Inability to understand and sign the informed consent form
* Known previous inability to perform spirometry
* Contraindications to perform spirometry as listed in the standardization of Spirometry 2019 update (Graham et al., 2019)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In principle, all patients with a spirometry indication diagnosis or monitoring of their airway disease of 16 years or older will be eligible for at-home spirometry.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Successful spirometry | 1 day: Participant will perform one spirometry session including several manoeuvres
  Occurrence (expressed as percentage of patients) of home spirometry being graded A, following technical standards of the American Thoracic Society (ATS) and the European Respiratory Society (ERS) (Graham, B. L. et al.)
Clinically useful spirometry | 1 day: Participant will perform one spirometry session including several manoeuvres
  Occurrence (expressed as percentage of patients) of home spirometry being graded A, B or C, following technical standards of the American Thoracic Society and the European Respiratory Society (Graham, B.L. et al.)

SECONDARY OUTCOMES:
Quality of spirometry, following ATS/ERS grading of spirometry | 1 day: Participant will perform one spirometry session including several manoeuvres
  Quality of spirometry performed as rated by the device application using the American Thoracic Society /European Respiratory Society (ERS) grading of spirometry on a scale from A (≥3 acceptable and repeatability within 0.150 litre) to F (zero acceptable or usable) (Graham, B. L. et al.)
Quality of spirometry curves as scored by independent spirometry professionals | 1 day: Participant will perform one spirometry session including several manoeuvres
  Quality as assessed by visual inspection of curves and values by two or three (in case of disagreement between the first two) independent spirometry professionals whether manoeuvres are acceptable or not
Healthcare professional's view on the added value of home spirometry | Immediately after completion of spirometry measurements
  Individual scores on a 5-points Likert-scale of questions asked to healthcare professionals regarding the added value of home spirometry for monitoring and diagnosing of asthma and COPD (the Likert-scales range from strongly disagree to strongly agree)
Patient's view on the added value of home spirometry | Immediately after completion of spirometry measurements
  Individual scores on a 5-points Likert-scale of questions asked to the patient on the benefit of home spirometry (the Likert-scales range from strongly disagree to strongly agree)
Degree of feasibility of home spirometry as rated by the healthcare professional | Immediately after completion of spirometry measurements
  Individual scores on a 5-points Likert-scale of questions on the feasibility of home spirometry, scored by health professionals, including four questions of a validated tool as published by Weiner et al.

OTHER OUTCOMES:
Agreement between Forced Expiratory Volume in the first second (FEV1) obtained from home spirometry and from spirometry assessed at the general practice | 1 week: participant is performing one home-spirometry session and within the same week one session at the general practice
  Mean difference (with 95% confidence interval) between the individual highest FEV1 value obtained from home spirometry and the FEV1 value from spirometry assessed at the general practice
Agreement between Forced Vital Capacity (FVC) obtained from home spirometry and from spirometry assessed at the general practice | 1 week: participant is performing one home-spirometry session and within the same week one session at the general practice
  Mean difference (with 95% confidence interval) between the individual highest FVC value obtained from home spirometry and the FVC value from spirometry assessed at the general practice
Occurrence of patients requiring video assistance by a spirometry professional | 1 day: Participant will perform one spirometry session including several manoeuvres
  Percentage of patients requiring assistance through a video connection with performing spirometry
Level of required assistance by a spirometry professional | 1 day: Participant will perform one spirometry session including several manoeuvres
  Mean total time in minutes spent per patient by a spirometry professional for performing home spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Janwillem Kocks, Principal Investigator — General Practitioners Research Institute
Locations (2):
- GPRI, Groningen, Netherlands
- Karolinska Institute, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459